CLINICAL TRIAL: NCT03222102
Title: Ventral Hernia Prevention After Liver Transplantation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the changed standard regarding access for liver transplantation, this no longer complied with the requirements of the study protocol.
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Ventral hernia prevention
Record Dates: First submitted 2017-07-17; First posted 2017-07-19 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Ventral Hernia; Liver Transplantation
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phasix mesh (Experimental): Phasix mesh will be affixed to the exposed fascia after closure of the Abdomen in the course of liver transplantation.
  Interventions: Device: Phasix mesh
- Standard surgery (No Intervention): Surgery will be performed according to routine, without the use of Phasix mesh.

INTERVENTIONS:
Device: Phasix mesh — After the closure of the Abdomen, Phasix mesh will be placed and affixed on the exposed fascia.
  Arms: Phasix mesh

SUMMARY:
This study aims to evaluate if the risk of developing ventral hernia after liver transplantation can be reduced through the prophylactic implantation of a synthetic, fully resorbable mesh "Phasix" in the course of liver transplantation.

Patients will be randomized in a 1:1 ratio to receive either Phasix mesh or standard surgery without the use of Phasix.

Ultra-sound examinations of the wound area will be performed 14 days, 3, 6 and 12 months after liver transplantation. Furthermore, presence of infections, seroma, pain and other problems in the wound area will be assessed.

DETAILED DESCRIPTION:
Ventral hernia is a frequently occurring complication following liver transplantation, with a reported risk in the literature ranging from 5% to 25%.

This study aims to evaluate if the risk of developing ventral hernia after liver transplantation can be reduced through the prophylactic implantation of a synthetic mesh "Phasix" in the course of liver transplantation.

PHASIX™ Mesh is a fully resorbable mesh implant prepared from poly-4-hydroxybutyrate (P4HB). Absorption of the mesh material occurs within 12 to 18 months.

Patients will be randomized in a 1:1 ratio to receive either Phasix mesh in the course of liver transplantation or standard surgery without the use of Phasix.

Ultra-sound examinations of the wound area will be performed 14 days, 3, 6 and 12 months after liver transplantation. Furthermore, presence of infections, seroma, pain and other problems in the wound area will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* First transplantation
* Signed Informed Consent

Exclusion Criteria:

* Combined transplantation
* Revisions after liver transplantation
* Patients who already received laparotomy or transverse upper laparotomy (longer than 15 cm)
* Preexisting abdominal wall hernia except umbilical hernia after liver transplantation
* Pregnant/lactating women
* Known allergies to tetracycline hydrochloride and kanamycin sulfate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2023-11-04 (Actual); Study Completion 2023-11-04 (Actual)

PRIMARY OUTCOMES:
Incidence of ventral hernia | 12 months after liver transplantation
  Evaluated by ultra-sound imaging

SECONDARY OUTCOMES:
Infections | 12 months after liver transplantation
  Number of infections in the wound area, assessed by clinical evaluation
Wound healing disorders | 12 months after liver transplantation
  Presence of wound healing disorders in the wound area, assessed by clinical evaluation
Seroma | 12 months after liver transplantation
  Presence of seroma in the wound area, assessed by clinical evaluation
Hematoma | 12 months after liver transplantation
  Number of hematoma in the wound area, assessed by clinical evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz; Klin. Abteilung für Transplantationschirurgie, Graz, Austria

IPD SHARING:
Plan to Share IPD: No